CLINICAL TRIAL: NCT03902197
Title: A Phase II Study of CD19 hsCAR-T for Refractory/Relapsed CD19+ B-ALL Patients Previously Treated With Cell Therapy
Brief Title: CD19 hsCAR-T for Refractory/Relapsed CD19+ B-ALL Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Beijing Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19hsCAR20190401
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-03

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: CD19 hsCAR-T; B-ALL; Humanized selective CAR
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 hsCAR-T (Experimental): This cohort will be administrated by T cells transduced with lentivirus vectors expressing CD19 hsCAR
  Interventions: Biological: CD19 hsCAR-T

INTERVENTIONS:
Biological: CD19 hsCAR-T — CD19 hsCAR-T will be administered by I.V. infusion

SUMMARY:
This Phase II study is to evaluate the efficacy and safety of a CD19-targeting humanized selective CAR-T (CD19 hsCAR-T) in refractory/relapsed CD19+ B-ALL leukemia patients who have no available curative treatment options, have a limited prognosis with currently available treatments, and were previously treated with a B cell directed cell therapy.

DETAILED DESCRIPTION:
CD19+ B-ALL patients who have relapsed after murine-based CD19 CAR-T (CD19mCAR-T) treatment and/or have limited clinical response to CD19mCAR-T will be enrolled to receive CD19 hsCAR-T treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with refractory/relapse B-cell ALL with no available curative treatment options (such as autologous or allogeneic SCT);
2. Subjects previously treated with B cell-directed engineered cell therapy are eligible if they meet the following criteria:

   1. relapsed and/or MRD-positive after prior cell therapy;
   2. partial response to prior cell therapy;
   3. Clinical and laboratory data are available;
3. Documented CD19 expression after previous B cell-directed therapies;
4. Aged 1 to 75 years;
5. KPS>40；
6. At least 2 weeks or 5 drug half-lives, whichever is shorter must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy;
7. Women of childbearing potential must have a urine pregnancy test taken and proven negative prior to the treatment. All patients agree to use reliable methods of contraception during the trial period and throughout the last follow-up visit;
8. Subjects with relapsed disease after prior allogeneic SCT (myeloablative or non-myeloablative) will be eligible if the patients do not present with active GVHD and are not undergoing immunosuppressive regimes;
9. Patients with CNS3 (WCB ≥5/mL in CSF with presence of lymphoblasts) disease will be eligible if the CNS disease is responsive to therapy;
10. Participation in the clinical trials should be voluntary with signed informed consent.

Exclusion Criteria:

1. Patients with hypervolemia (white blood cell count> 50 x 10^9 / L) or rapidly progressive disease that in the estimation of the investigators and sponsors would compromise the patient's ability to complete the study;
2. History of melanoma skin cancer or other primary tumors (eg, cervical cancer, bladder cancer, breast cancer) (except for those with 3 years or longer of cure);
3. Patients with fungal, bacterial, viral, or other uncontrollable infections or infections requiring Level 4 isolation (UTI or inoculation assays may be performed if necessary);
4. Patients with positive results for HIV, HBV, HCV tests;
5. With CNS disorders such as cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or autoimmune disease with CNS involvement;
6. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac diseases within 12 months of enrollment, or with cardiac atrial or cardiac ventricular lymphoma;
7. Patients that are receiving anticoagulant therapy or have ever coagulation disorders;
8. Any medical condition that in the judgment of the sponsors/investigators is likely to interfere with assessment of safety or efficacy of study;
9. History of severe immediate hypersensitivity reaction to any of the agents used in this study;
10. Female patients who are pregnant or breastfeeding;
11. Feasibility assessment during screening demonstrates <30% transduction of target lymphocytes, or insufficient expansion (< 5-fold) in response to CD3/CD28 co-stimulation;
12. Patients with any uncontrolled diseases that are unsuitable for enrollment;
13. CNS3 disease that is progressive on therapy, or with CNS parenchymal lesions that might increase the risk of CNS toxicity;
14. Any situation that is considered to potentially increase the risk of the subject or interfere with the outcome of the study;
15. Patients who have been enrolled in other clinical studies.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-22 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) within 3 months | 3 months
  Overall response rate (ORR) within 3 months after infusion of CD19 hsCAR-T

SECONDARY OUTCOMES:
Best overall response (BOR) | 3 months
  Best overall response (BOR) of complete remission (CR) or CR with incomplete blood count recovery (CRi) within 3 months after CD19 hsCAR-T infusion
Duration of remission (DoR) | 1 year
  Duration of remission (DoR) within 1 year after CD19 hsCAR-T infusion (Duration of remission (DOR) is defined as the duration from the date when the response criteria of CR or CRi is first met to the date of relapse or death due to ALL)
Event free survival within 1 year | 1 year
  Event free survival within 1 year (Event free survival is defined as the time from start of the first infusion to the earliest of death from any cause or relapse)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | 6 months
  Safety and tolerability of CD19 hsCAR-T: frequency and severity of adverse events, including, but not limited to, cytokine release syndrome (CRS) and macrophage activation syndrome (MAS)

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Chen, PhD, Principal Investigator — Xuanwu Hospital, Beijing; Huyong Zheng, MD, PhD, Principal Investigator — Beijing Children's Hospital
Locations (2):
- China (2):
  - Beijing Children's Hospital Capital Meidcal University, Beijing, Beijing Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality